CLINICAL TRIAL: NCT06159881
Title: Customized Crosslinking: Safety and Efficacy in an Epithelium-off Accelerated-pulsated Protocol for Thin Keratoconus Corneas
Brief Title: Customized Crosslinking: Safety and Efficacy in an Epithelium-off Accelerated-pulsated Protocol for Thin Keratoconus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17 CI 09 015 008
Record Dates: First submitted 2023-11-28; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Keratoconus
Keywords: Progression; Customized; Cross-Linking
MeSH Terms: conditions — Keratoconus; Disease Progression | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized cross linking (Experimental): Participants were treated with personalized energy cross linking according to their thinnest point corneal pachymetry
  Interventions: Procedure: Corneal Cross Linking

INTERVENTIONS:
Procedure: Corneal Cross Linking — Total fluence adapted to thinnest point pachymetry

SUMMARY:
The goal of this clinical trial is to document corneal ectasia stability in patients with keratoconus diagnosis treated with personalized cross linking energy. The main questions it aims to answer are:

* Is it effective while using personalized (reduced) energy?
* Is it safe for corneas thinner than 400 microns? Participants will be treated with personalized energy corneal cross linking and posteriorly, will attend subsequent follow-up consults

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus diagnosed with corneal tomography/topography
* Thinnest point pachymetry below 400 microns

Exclusion Criteria:

* Previous corneal cross linking history
* Corneal scars not allowing best corrected visual acuity of 20/100 or better
* Previous corneal hydrops history
* Psychomotor retardation history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Keratometry stability | Baseline and 6 months
  Stability documented by changes in keratometries (measured in diopters) obtained with corneal tomography, as well as uncorrected visual acuity observed in follow up consults
Pachymetry stability | Baseline and 6 months
  Stability documented by changes in pachymetry (measured in microns) obtained with corneal tomography
Uncorrected visual acuity stability | Baseline, 72 hours, 1 week, 3 months and 6 months
  Stability documented by changes in uncorrected visual acuity (measured in logarithm of the minimum angle of resolution) obtained on physical examiantion
Corneal endothelium safety | Baseline, 72 hours, 1 week, 3 months and 6 months
  Corneal endothelial cell count obtained by specular microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Graue, MD, MSc, Study Director — Instituto de Oftalmología Conde de Valenciana
Locations (1):
- Instituto de Oftalmología Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hafezi F, Kling S, Gilardoni F, Hafezi N, Hillen M, Abrishamchi R, Gomes JAP, Mazzotta C, Randleman JB, Torres-Netto EA. Individualized Corneal Cross-linking With Riboflavin and UV-A in Ultrathin Corneas: The Sub400 Protocol. Am J Ophthalmol. 2021 Apr;224:133-142. doi: 10.1016/j.ajo.2020.12.011. Epub 2021 Jan 30. PMID 33340508
- [Background] Lang PZ, Hafezi NL, Khandelwal SS, Torres-Netto EA, Hafezi F, Randleman JB. Comparative Functional Outcomes After Corneal Crosslinking Using Standard, Accelerated, and Accelerated With Higher Total Fluence Protocols. Cornea. 2019 Apr;38(4):433-441. doi: 10.1097/ICO.0000000000001878. PMID 30681515
- [Background] Nath S, Shen C, Koziarz A, Banfield L, Nowrouzi-Kia B, Fava MA, Hodge WG. Transepithelial versus Epithelium-off Corneal Collagen Cross-linking for Corneal Ectasia: A Systematic Review and Meta-analysis. Ophthalmology. 2021 Aug;128(8):1150-1160. doi: 10.1016/j.ophtha.2020.12.023. Epub 2020 Dec 28. PMID 33383093